CLINICAL TRIAL: NCT03587285
Title: A Pilot Study of Hormonal Therapy Combined With Central Memory T Cells (Tcm) for Patients With Advanced Prostate Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Songtao Xiang, MD, PhD, Guangzhou University of Traditional Chinese Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2017-05-01
Record Dates: First submitted 2018-07-03; First posted 2018-07-16 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Prostatic Neoplasms
Keywords: prostate cancer; central memory T cell
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): metastatic hormone-sensitive prostate cancer (mHSPC):After diagnosis of mHSPC, patients receive infusions of autologous Tcm cells intravenously on Day 1 and Day 42, followed by hormonal therapy of maximal androgen blockade (LHRH-a + Anti-androgen).
  Interventions: Biological: Tcm+ Goserelin acetate+ Bicalutamide
- Arm 2 (Experimental): metastatic castration-resistant prostate cancer (mCRPC):After diagnosis of mCRPC, patients receive infusions of autologous Tcm cells intravenously on Day 1 and Day 42, followed by goserelin acetate monthly. Abiraterone acetate 1000 mg orally daily plus prednisone 5 mg orally twice daily will be also administered continuously during the duration of the trial.
  Interventions: Biological: Tcm+Goserelin acetate+Abiraterone acetate

INTERVENTIONS:
Biological: Tcm+ Goserelin acetate+ Bicalutamide — Autologous Tcm cells administered intravenously on Day 1 and Day 42,3.6mg goserelin acetate injection administered subcutaneously monthly,50 mg bicalutamide administered orally daily
  Arms: Arm 1
Biological: Tcm+Goserelin acetate+Abiraterone acetate — Tcm cells administered intravenously on Day 1 and Day 42,3.6mg goserelin acetate injection administered subcutaneously monthly,1000 mg abiraterone acetate administered orally daily plus 5 mg prednisone administered orally twice daily
  Arms: Arm 2

SUMMARY:
The purpose of this study is to evaluate the feasibility, safety and oncological efficacy of hormonal therapy combined with autologous Tcm cells for patients with advanced prostate cancer.

DETAILED DESCRIPTION:
Adoptive cancer immunotherapy,the infusion of tumor-reactive T cells to patients,represents a promising approach for the treatment of advanced metastatic disease.It has been shown that central memory T cells (Tcm) were the optimal antitumor T cells for adoptive cell transfer in cancer patients.However,the potential of autologous Tcm cells to treat the advanced prostate cancer has not been evaluated.

This is an open-label pilot study to determine if the infusion of autologous Tcm cells combined with hormonal therapy is safe and effective for the treatment of advanced prostate cancer.This study will have the following two cohorts:Cohort A) metastatic hormone-sensitive prostate cancer (mHSPC) treated with maximal androgen blockade plus autologous Tcm cells and Cohort B) metastatic castration-resistant prostate cancer (mCRPC) treated with abiraterone acetate plus autologous Tcm cells.A total of 60 evaluable subjects will be enrolled over an enrollment period of 24 months.The study is planned to enroll approximately 30 evaluable subjects in each treatment cohort.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who understand and sign the consent form for this study
* Males age ≥18 years
* Subjects diagnosed with metastatic hormone-sensitive prostate cancers (mHSPC) or metastatic castration-resistant prostate cancer (mCRPC)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Expected survival time of at least 24 months
* Adequate hematologic, renal, and liver function: WBC greater than 3.5 x 109/L; Absolute neutrophils count greater than 1.5 x 109/L; Platelet count greater than 80 x 109/L; Hemoglobin at least 90g/L; AST less than 2 x upper limit of normal (ULN); Creatinine less than 1.5 x ULN
* No obvious abnormalities in the electrocardiogram

Exclusion Criteria:

* Clinically significant cardiovascular disease: New York Heart Association (NYHA) class III or IV chronic congestive heart failure, coronary heart disease (myocardial infarction within 6 months); cardiac arrhythmia requiring anti-arrhythmic drug (beta-blocker or digoxin is allowed to be used); uncontrolled high blood pressure
* HIV infection
* Acute exacerbation of chronic hepatitis A or hepatitis B infection
* The subject has uncontrollable seizures required pharmacotherapy (such as steroids or antiepileptic drugs)
* The subject has a history of allogeneic organ transplants
* Subject with irregular hemorrhagic disease
* The subject receives dialysis treatment The subject has a history of other malignant tumor except subjects with curable basal cell carcinoma, superficial bladder tumor or other tumors has been cured over three years of study entry
* The subject has a history of gastrointestinal hemorrhage within 30 days of study entry
* The subject has an allergic history or is allergic to the drug in this study
* The subject has serious diseases of respiratory, nervous or mental system
* Subject with immune disease, auto-immune disease requires systemic ongoing immunosuppressive therapy
* The subject has problems with drug or alcohol abuse
* Major surgery within 4 weeks of enrollment
* Prior autologous bone marrow transplantation within 4 weeks of enrollment
* The subject has participated in any other therapeutic clinical trial with an experimental drug in the 4 weeks prior to this trial
* The subject has any other unsuitable or adverse condition to be determined by the investigator
* Any medical intervention or any circumstances that could compromise the safety and compliance of the trial subjects

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-09-23 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidences of adverse events or serious adverse events (AE and SAE) | 2 years
  This is graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) grading scale, version 4.0

SECONDARY OUTCOMES:
Time to castration-resistance (TCR) in mHSPC patients | 2 years
  Defined as the time from treatment initiation to the first castration-resistant event (radiographic disease progression, prostate-specific antigen (PSA) progression or the occurrence of the first symptomatic skeletal event), whichever occurs first
Overall survival (OS) | 2 years
  Defined as time from treatment initiation to death
Progression-free survival (PFS) | 2 years
  Defined as the time from treatment initiation to disease progression, relapse or death due to any cause, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Songtao Xiang, MD, Principal Investigator — Guangzhou University of Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Chinese Medicine, Guangzhou University of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided